CLINICAL TRIAL: NCT07123870
Title: Effect of Combined Intravenous-Inhalational Anesthesia (CIVIA) on Postoperative Recovery Patterns.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Yuksek, Clinical Professor, Kocaeli City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAEK/10.bI.02
Record Dates: First submitted 2025-07-28; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Recovery; Inhalation Anesthesia; Total Intravenous Anesthesia
Keywords: CIVIA; TIVA; sevoflurane; desflurane; postoperative recovery
MeSH Terms: interventions — Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant: The participant will be unaware of which anesthesia method is involved in the perioperative period.
  Care Provider: The second anesthesiologist is responsible for the patient's recovery after the anesthesia is terminated and will be unaware of which anesthetic method was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sevoflurane combined with TIVA (Experimental): Combined anesthesia with sevoflurane and intravenous agents. A 0.5 MAC sevoflurane combined with TIVA. TIVA will be administered using target-controlled infusion (TCI) with the Eleveld pharmacokinetic model, utilizing a propofol-remifentanil combination, and guided by BIS monitoring.
  Interventions: Drug: Sevofluorane
- Desflurane combined with TIVA (Experimental): Combined anesthesia with desflurane + intravenous agents. TIVA will be administered using target-controlled infusion (TCI) with the Eleveld pharmacokinetic model, utilizing a propofol-remifentanil combination, and guided by BIS monitoring. Efect site concentration will be aimed for TIVA
  Interventions: Drug: Desflurane
- TIVA (Experimental): Total Intravenous Anesthesia. TIVA will be administered using target-controlled infusion (TCI) with the Eleveld pharmacokinetic model, utilizing a propofol-remifentanil combination, and guided by BIS monitoring. Efect Site concentration will be aimed. for sole TIVA, 2-4mcg/ml propofol and 1-4ng/ml remifentanil will bu used according to BIS monitoring. 40-60 range will be used for BIS.
  Interventions: Drug: Total Intravenous Anesthesia(TIVA)

INTERVENTIONS:
Drug: Sevofluorane — In this group of patients, <0.5 MAC sevoflurane will be used in combination with TIVA. (TIVA method described above)
  Other Names: Sevoflurane Combined Anesthesia
  Arms: Sevoflurane combined with TIVA
Drug: Desflurane — In this group of patients, <0.5 MAC Desflurane will be used in combination with TIVA.
  Other Names: Desflurane Combined anesthesia
  Arms: Desflurane combined with TIVA
Drug: Total Intravenous Anesthesia(TIVA) — In this group, TIVA will be applied with the combination of BIS-guided propofol + remifentanil.
  Other Names: Total Intravenous Anesthesia
  Arms: TIVA

SUMMARY:
This study was planned as a single-center, prospective, randomized trial. Adult patients undergoing elective spinal surgery lasting longer than three hours, performed in a neurosurgery operating room, will be evaluated. Patients managed with three different anesthesia methods currently used will be examined for recovery patterns:

1. Total intravenous anesthesia (TIVA),
2. TIVA Combined anesthesia with sevoflurane and intravenous agents (sevoflurane-CIVIA),
3. TIVA Combined anesthesia with desflurane and intravenous agents (desflurane-CIVIA).

Recovery patterns include; extubation time, eye opening time, emergence agitation, postoperative nausia and vomiting and postoperative recovery unit discharge time.

DETAILED DESCRIPTION:
The aim of this study was to compare the effects of different anesthesia methods applied in spinal surgeries lasting longer than three hours on postoperative recovery time. Specifically, it aimed to determine the contribution of low-dose (0.5 MAC) desflurane or sevoflurane combined intravenous anesthesia (CIVIA) approaches compared to total intravenous anesthesia (TIVA) on recovery parameters such as patient recovery time, extubation time, and time to consciousness. It also aimed to investigate whether the desflurane-containing combination resulted in a faster recovery than the sevoflurane-containing combination.

TIVA will be administered using target-controlled infusion (TCI) with the Eleveld pharmacokinetic efect site model, utilizing a propofol-remifentanil combination, and guided by BIS monitoring.

Outputs:

Eye opening time (the time from the end of anesthesia until the patient's eye opening for verbal stimuli) Extubation time (the time from the end of anesthesia until extubation) Richardson agitation sedation and RAMSEY scale values, and Emergence agitation incidence.

Postoperative nausea and vomiting incidence (PONV). Time to discharge from the PACU and time to an Aldrate score >9 will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for spine surgery
* Expected surgery duration longer than 3 hours
* Use of intraoperative neuromonitoring
* BIS-guided anesthesia administered
* TIVA (with TCI) as the primary anesthetic technique
* Age >18 years

Exclusion Criteria:

* Emergency surgeries
* Patients receiving sole inhaled anesthesia (no TIVA)
* Perioperative dural injury
* Intraoperative severe hypotension requiring inotropic support
* Hypothermia (based on temperature measured before recovery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Extubation time | First postoperative hour
  Extubation time in patients after all anesthetic drugs have been discontinued

SECONDARY OUTCOMES:
Eye opening | First postoperative hour
  time brtween anesthesia terminated and aye opening after surgery

OTHER OUTCOMES:
Richmond Agitation-Sedation Scale (RASS) | first 2 hours postoperatively
  Richmond Agitation-Sedation Scale (RASS) A 10-point scale ranging from +4 (combative) to -5 (unarousable). Measures agitation, sedation level, and responsiveness. Helps guide sedation management and assess recovery from anesthesia.
Postoperative Nausia and Vomiting | First 2 postoperative hours
  Postoperative Nausia and Vomitting incidance
PACU discharge time | First 2 postoperative hours
  The time between the termination of anesthesia and the patient being discharged from the postoperative recovery room (PACU) with an Aldrete score of >9. It is calculated in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YUKSEK, Md, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmıt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolf A, Selpien H, Haberl H, Unterberg M. Does a combined intravenous-volatile anesthesia offer advantages compared to an intravenous or volatile anesthesia alone: a systematic review and meta-analysis. BMC Anesthesiol. 2021 Feb 15;21(1):52. doi: 10.1186/s12871-021-01273-1. PMID 33588751
- [Background] Song T, Wu LJ, Li L. Comparison of combined intravenous and inhalation anesthesia and total intravenous anesthesia in laparoscopic surgery and the identification of predictive factors influencing the delayed recovery of neurocognitive function. Front Med (Lausanne). 2024 Mar 25;11:1353502. doi: 10.3389/fmed.2024.1353502. eCollection 2024. PMID 38590312
- [Background] Wang Y, Cao M, Cao G, Liu Y, Zhang Y. Effect of combined intravenous-inhalation anesthesia on postoperative cognitive dysfunction after laparoscopic radical resection of cervical cancer: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Nov 6;99(45):e23124. doi: 10.1097/MD.0000000000023124. PMID 33157991